CLINICAL TRIAL: NCT06452199
Title: The BEGIN Study Bifidobacterium Infantis to Newborns: Effects of Modulating the Gut Microbial Composition on Growth, Immune Function and Inflammatory Conditions
Brief Title: The BEGIN Study Bifidobacterium Infantis to Newborns: Effects of Modulating the Gut Microbial Composition on Growth, Immune Function and Inflammatory Conditions - a Randomized Placebo-controlled Double-blinded Intervention Trial
Acronym: BEGIN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other); Gødstrup Hospital (Other); Regionshospitalet Horsens (Other); Technical University of Denmark (Other); Statens Serum Institut (Other); University of Copenhagen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: BEGIN 2024
Record Dates: First submitted 2024-05-22; First posted 2024-06-11 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-04

CONDITIONS: Healthy; Healthy Nutrition
Keywords: Microbiota; Gastrointestinal Microbiome; Probiotics; Bifidobacterium longum subspecies infantis; Paediatrics; Infant; Child; Immunology; Infections; Inflammation; Growth and Development; Colic; Respiratory Tract Diseases; Metabolism
MeSH Terms: conditions — Infections; Inflammation; Colic; Respiratory Tract Diseases

STUDY DESIGN:
Intervention Model Description: Randomised controlled double-blinded intervention trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- B. infantis (Active Comparator): The investigational product to be tested is a Probio-Tec® I Stick-0.16 IF, containing 1.0 g of a standardized fine powder consisting of a food constituent, the freeze-dried culture of Bifidobacterium longum subsp. infantis Bifin02 (DSM33361).
  The infant dietary supplement is supposed to be mixed with a little human milk or clean water.
  Interventions: Dietary Supplement: B. infantis
- Placebo (Placebo Comparator): Identical looking placebo.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: B. infantis — 1000 newborn children are randomized 50/50 to receive either B. infanits or placebo in a dietary supplement, for daily oral administration in three weeks from 7 days of age.
  Other Names: Bifidobacterium longum subsp. infantis Bifin02 (DSM33361)
  Arms: B. infantis
Dietary Supplement: Placebo — Identical looking placebo (without any probiotics/B. infantis) for double-blinded daily oral administration in three weeks from 7 days of age.
  Arms: Placebo

SUMMARY:
The goal of The BEGIN Study, a randomized controlled double-blinded intervention trial, is to learn if probiotics, with Bifidobacterium longum subspecies infantis Bifin02 (B. infantis), given to healthy newborns can affect various health outcomes and to explore impacts of the infant gastrointestinal microbiome. The main questions it aims to answer are:

* Does B. infantis probiotics impact immune function and does it lower the number of bacterial infections and use of antibiotics?
* Does B. infantis probiotics impact overall health, development, growth and wellbeing?
* Does B. infantis probiotics impact inflammatory diseases, allergies and autoimmune diseases

Researchers will compare B. infantis probiotics to a placebo (a look-alike substance that contains no probiotic) to see if B. infantis colonization impact the human immunesystem and various clinical and biochemical health markers.

Participants (parents) will

* Orally administrate the B. infantis probiotic to their newborn child daily in three weeks from 7 days of age.
* Answer baseline and follow up questionnaires in a study app
* Take five stool samples from the child and one stool sample from the mother
* Collect a 4 week of passive dust sample at home (Electrostatic Dust fall Collector)
* Donate one dried bloodspot and one blood sample from their child

ELIGIBILITY:
Inclusion Criteria:

* Infants born at term (above gestational week 37)
* Infants born in Region Midtjylland Denmark receiving a Danish CPR number.
* Parents age is above 18
* At least one parent holds a smartphone (for study app) and is able to fill out Danish questionaries
* Both legal parents are willing and able to provide written informed consent prior to participation, regarding both themselves and their future child.

Exclusion Criteria:

* Multiple pregnancy
* Child diagnosed with immune deficiency, renal, gastrointestinal, hepatic, or endocrine diseases
* Parents expecting to give other probiotics

Ages: 1 Day to 7 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1000 (Estimated)
Dates: Start 2024-06-10 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2043-11 (Estimated)

PRIMARY OUTCOMES:
Prescriptions of antibiotics | First assessment at 1 year and up to 18 years follow-up
  Number of prescriptions of antibiotics among participants, as a measure of bacterial infections.

SECONDARY OUTCOMES:
The intestinal microbiota and B. infantis colonization | 1 year
  Stool samples collected during the first year of life and tested with shutgun metagenomics, assessing the microbial composition..
Antibiotic resistance genes (ARGs) | 1 year
  Amount of Antibiotic resistance genes (ARGs) in participants microbial community in stool samples. Identification with shutgun metagenomics. Assessing the microbial composition and diversity.
Colic | 3 months
  Parents' observations registered in study app. Duration of crying in the first three months of life. Defined as Wessels criteria:
  Crying for three or more hours a day, three or more days a week, for three or more weeks.
Bowel function, stool consistency | 3 months
  Parents' observations registered in study app, related to their infant child's stool consistency measured at the Infant Stool Scale
Bowel function, stool frequency. | 3 months
  Parents' observations of their infant child's frequency of stool passings, registered in study app
Bowel function, laxatives | 3 months
  Parents' reported use of medical laxatives for their infant child, registered in study app and reported as amount of days using the laxative.
High sensitive C-reactive protein (hs-CRP) | 1 year
  Blood biomarker: Low-grade systemic inflammation. Unit of measurement: mg/l
Cluster of Differentiation 163" (CD163) | 1 year
  Blood biomarker: Macrophage-mediated inflammation and insulin-sensitivity. Unit of measurement: mg/l
Plasma Calprotectin | 1 year
  Blood biomarker: Intestinal inflammation. Unit of measurement: µg/l
Allergies, Immunoglobulin E (IgE) | 1 year
  Blood marker: Allergies. Specific IgE against the 11 most common inhalation allergens and IgE directed against Egg white, cow's milk, codfish, wheat, peanut and soybean. Unit of measurement: IU/l
Allergies | 1 year
  Self reported allergy symptoms
Growth, weight gain | First assessment at 1 year and up to 18 years follow-up
  Measured as weight gain in kilograms
Growth | First assessment at 1 year and up to 18 years follow-up
  Growth velocity and weight-for-length z-scores, measured in kilograms and centimeters and combined for Z-scores.
Growth, IGF-1 (Insulin-like Growth Factor-1) | 1 year
  Blood biomarker: Mediating the growth-promoting effects of growth hormone. Unit of measurement: µg/l
Body composition | 3 months
  Measured by air displacement plethysmography (ADP) (Pea Pod) estimating body fat
Body composition | 3 months
  Measured by air displacement plethysmography (ADP) (Pea Pod) estimating muscle mass.

OTHER OUTCOMES:
Hospital admissions | First assessment at 1 year and up to 18 years follow-up
  Number of hospital admissions. Registered at Landspatientregistret
Febrile episodes | 1 year
  Number of days with a fever during the last month. A febrile episode is characterized as a body temperature at 38 degrees Celsius or above. Self-reported in a monthly questionnaire in study app.
Asthma Control Test | 1 year, possible later follow-up
  Participants reporting symptoms of astma or astmatic bronkitis, will be asked to complete the Asthma Control Test. The scores range from 5 (poor control of asthma) to 25 (complete control of asthma), with higher scores reflecting greater asthma control. An ACT score >19 indicates well-controlled asthma.
Asthmatic Bronchitis, prescriptions | First assessment at 1 year
  Number of prescriptions of medicine for asthmatic bronchitis; Ventoline, Airomir, Flixotide, Aerobec, Montelukast / Singulair.
Asthmatic bronchitis, hospitalization | First assessment at 1 year
  Number of hospitalizations due to asthmatic bronchitis.
Diaper rash | 1 year
  Atopic skin symptoms in diaper area. Self-reported by the childs parents as affected red skin, distribution in centimeters .
Rhinoconjunctivitis | 1 year
  Measured as Mini Rhinoconjunctivitis quality of life questionnaire Mini RQLQ, adjusted to infants. 14 questions in five domains (activity limitation, practical problems, nose symptoms, eye symptoms, and non-nose/ eye symptoms), scores for each question is ranging from 0 to 6, with 0 reflecting no affection and 6 reflecting maximum affection.
Obesity | 18 years
  Measured as number of participants diagnosed with Obesity
Metabolic syndrome | 18 years
  Measured as number of participants diagnosed with Metabolic syndrome
Diabetes | 18 years
  Measured as number of participants diagnosed with Diabetes
Inflammatory bowel disease | 18 years
  Measured as number of participants diagnosed with of Morbus Crohn and/or Colitis Ulcerosa.
Dried blood spot for metabolomics | 3 months and 1 year
  The metabolomic method measures and compares large numbers of metabolites (for example shot chained fatty acids) present in the dried blood sample.
Bloodsample analyzed with Singlecell PBMC method | 1 year
  Single cell sequencing is a method profiling the peripheral blood mononuclear cells (PBMC), by isolating memory B, T and B-cells
Child stool sample | 1 year
  Stool samples collected at week 1, 4, 13, 28 and 52 will by qPCR or shutgun metagenomics examine the gut microbiome.
Mother stool sample | 1 month
  A stool sample from the pregnant mother, preferably prior to or during birth. To analyze mothers microbial colonization, that may be transferred to the child, e.g during vaginal birth.
Mother HMO-secretor status | 1 month
  The type of Human Milk Oligosaccharides (HMO) section in mothers' breastmilk, will be determined to exploratively study the relationship between types of HMO's, mothers HMO-secretor status and effects of B.infantis.
Asthma | up to 18 years follow-up
  Number of participants with prescriptions of medicine for asthma
Atopic disease (adjusted SCORAD grading) | First assessment at 1 year
  Atopic symptoms, eczema, registered in study-app with description of episodes of atopic dermatitis (adjusted SCORAD grading). Disease intensity is calculated based on six characteristics: erythema, edema, oozing/crusts, excoriations, lichenification, and dryness. Each characteristic is given a score between 0 and 3, where 0 is absent and 3 is severe. The scores for each characteristic are added together for a total intensity score of up to 18.
Atopic disease, local steroids | First assessment at 1 year and up to 18 years follow-up
  Number of participants with prescriptions of local steroids to treat eczema.

CONTACTS AND LOCATIONS:
Overall Officials: Sune Rubak, MD, Phd, Principal Investigator — Department of Paediatrics, Aarhus University Hospital (AUH) and Aarhus University; Kurt Kristensen, MD, Phd, Principal Investigator — Steno Diabetes Centre Aarhus and Department of Paediatrics (AUH) and and Aarhus University
Locations (2):
- Denmark (2):
  - Regional Hospital Gødstrup, Herning, Central Jutland
  - Regional Hospital Horsens, Horsens, Central Jutland

IPD SHARING:
Plan to Share IPD: Yes
Anonymized data that underlie the results reported in study articles (text, tables, figures, and appendices).
  The laws related to the handling of personal data will be followed and results are processed in accordance with the General Data Protection Regulation (GDPR) and the Danish Data Protection Act (Databeskyttelsesforordningen and Databeskyttelsesloven).
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After the study has been finalized
Access Criteria: Researchers who provide a methodologically sound proposal.

REFERENCES:
- See also: studywebsite for participants — http://www.beginstudy.dk